CLINICAL TRIAL: NCT02632266
Title: Effect of Extensively Hydrolyzed Liquid Human Milk Fortifier on Growth and Tolerance in Moderately Premature Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00002292
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Complication of Prematurity
Keywords: prematurity; growth; nutrition; human milk fortifier
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Powder HMF (Active Comparator): Once patient has reached 80ml/kg/day of enteral feedings, 1 pack of powder HMF will be added to 50 ml of human or donor breast milk, then increased to a maximum of 2 packs for 50 ml following the unit feeding advancement protocol and this will be continued up until 48 hours prior to discharge.
  Interventions: Dietary Supplement: Powder HMF
- Liquid HMF (Active Comparator): Once patient has reached 80ml/kg/day of enteral feedings, researchers will add 1 packet (5 ml) of liquid HMF to 50 ml of human or donor breast milk, then increase to 2 packs to 50 ml following the unit feeding protocol and this will be continued up until 48 hours prior to discharge.
  Interventions: Dietary Supplement: Liquid HMF

INTERVENTIONS:
Dietary Supplement: Powder HMF — powder human milk fortifier
  Arms: Powder HMF
Dietary Supplement: Liquid HMF — Liquid human milk fortifier
  Arms: Liquid HMF

SUMMARY:
The purpose of this study is for the researchers to examine the safety and efficacy of liquid human milk fortifier (HMF) in moderately preterm infants compared to powdered human milk fortifier.

DETAILED DESCRIPTION:
This is a prospective, randomize, double-blinded study in preterm infants born between 28-34 weeks gestation admitted to the NICU at the University of Kansas Hospital. After obtaining informed consent, babies will be randomized to either liquid or powdered HMF using opaque, sealed envelopes with preassigned randomization. The feeding protocol as established in the KU NICU will be followed, beginning with initiation of trophic feeds, and advancement of enteral feeds depending on the gestational age and preceding illnesses. Once infants reach 80ml/kg/day of enteral feeds, human milk will be fortified to 22 kilocalories by adding either liquid or powdered fortifier. The beginning of the study(Study day 1) will be defined as reaching and tolerating 100ml/kg/day of 24 kilocalorie human milk fortified with either liquid or powdered fortifier. Enteral feeds will be advanced per unit protocol until they reach 150-160ml/kg/day and 110-120 kcal/kg/day. the volume of feeds will be adjusted based on the documented weight to provide energy and protein requirements as recommended by the ESPGHAN guidelines. Babies will be followed up until the time of NICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Inborn preterm infants born between 28 0/7 and 34 0/7 weeks gestation and fed either mother's own milk or donor human milk

Exclusion Criteria:

* Newborn infants <28 weeks and >34 weeks gestation, those with life threatening illness, congenital and chromosomal anomalies, gastrointestinal anomalies or necrotizing enterocolitis and fed premature formula

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Cumulative weight gain | Baseline to 36 Weeks post-conceptional age or Study Day 28, whichever is earlier
  Weight gain of baby during the course of the study
Change in weight | Baseline to 36 Weeks post-conceptional age or Study Day 28, whichever is earlier
  Weight gain of baby week-to-week, during the course of the study
Linear length | Baseline to 36 Weeks post-conceptional age or Study Day 28, whichever is earlier
  change in length week-to-week during the course of the study
Head growth | Baseline to 36 Weeks post-conceptional age or Study Day 28, whichever is earlier
  Change in head measurements week-to-week during the course of the study

SECONDARY OUTCOMES:
Nutrition biomarkers | Baseline to 36 Weeks post-conceptional age or Study Day 28, whichever is earlier
  Measurements of a baby's Ca, P, Mg, Alkaline Phosphatase and Prealbumin will be taken
Tolerance to enteral feeds | Baseline to 36 Weeks post-conceptional age or Study Day 28, whichever is earlier
  number of significant residuals, number of times feeds were held, NEC

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Pandey, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hylander MA, Strobino DM, Dhanireddy R. Human milk feedings and infection among very low birth weight infants. Pediatrics. 1998 Sep;102(3):E38. doi: 10.1542/peds.102.3.e38. PMID 9724686
- [Result] Lucas A, Cole TJ. Breast milk and neonatal necrotising enterocolitis. Lancet. 1990 Dec 22-29;336(8730):1519-23. doi: 10.1016/0140-6736(90)93304-8. PMID 1979363
- [Result] Greer FR, McCormick A. Improved bone mineralization and growth in premature infants fed fortified own mother's milk. J Pediatr. 1988 Jun;112(6):961-9. doi: 10.1016/s0022-3476(88)80227-0. PMID 3373407
- [Result] Cibulskis CC, Armbrecht ES. Association of metabolic acidosis with bovine milk-based human milk fortifiers. J Perinatol. 2015 Feb;35(2):115-9. doi: 10.1038/jp.2014.143. Epub 2014 Aug 7. PMID 25102321
- [Result] Thoene M, Hanson C, Lyden E, Dugick L, Ruybal L, Anderson-Berry A. Comparison of the effect of two human milk fortifiers on clinical outcomes in premature infants. Nutrients. 2014 Jan 3;6(1):261-75. doi: 10.3390/nu6010261. PMID 24394538
- [Result] Agostoni C, Buonocore G, Carnielli VP, De Curtis M, Darmaun D, Decsi T, Domellof M, Embleton ND, Fusch C, Genzel-Boroviczeny O, Goulet O, Kalhan SC, Kolacek S, Koletzko B, Lapillonne A, Mihatsch W, Moreno L, Neu J, Poindexter B, Puntis J, Putet G, Rigo J, Riskin A, Salle B, Sauer P, Shamir R, Szajewska H, Thureen P, Turck D, van Goudoever JB, Ziegler EE; ESPGHAN Committee on Nutrition. Enteral nutrient supply for preterm infants: commentary from the European Society of Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2010 Jan;50(1):85-91. doi: 10.1097/MPG.0b013e3181adaee0. PMID 19881390